CLINICAL TRIAL: NCT01035281
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Assignment, Efficacy Study of Nabilone in the Treatment of Diabetic Peripheral Neuropathic Pain
Brief Title: Efficacy Study of Nabilone in the Treatment of Diabetic Peripheral Neuropathic Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Valeant Canada, Valeant Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U Calgary # UCNABDPN01
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Diabetic Neuropathies
Keywords: Diabetic Neuropathies; Neuropathic Pain; Cannabinoids; Tree Number C10.668.829.300
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nabilone (Experimental): A one-week screening period will occur, during which pain scores and sleep scores will be tabulated. Following screening, a 4-week period of single blind treatment with flexible dosing of nabilone at 0.5 - 4 mg/day will initiate.
  Interventions: Drug: Nabilone, flexible dosing
- Placebo (Placebo Comparator): All subjects who experience at least a 30% reduction in their weekly mean pain score during the single blind flexible dosing phase will be considered a responder, and will be further continued in the study. During the double-blind portion of the study, subjects randomized to nabilone will continue on the dose of nabilone achieved at the completion of the single-blind phase, and this dose will be maintained throughout the double-blind phase. Subjects randomized to placebo will receive 1 mg of nabilone daily for one week, followed by 4 consecutive weeks of placebo. This dose of nabilone will permit a tapering for those subjects achieving a higher daily dose of nabilone during the single-blind phase, or will maintain those who were taking only 1 mg per day in the single-blind phase, preventing an abrupt termination of treatment in subjects who are randomized into the placebo portion.
  Interventions: Drug: Nabilone, flexible dosing

INTERVENTIONS:
Drug: Nabilone, flexible dosing — nabilone at 0.5 - 4 mg/day
  Other Names: Cesamet

SUMMARY:
Neuropathic pain occurs as a result of damage or disease of the peripheral or central nervous system. Regardless of its cause, neuropathic pain (NeP) leads to a characteristic clinical picture characterized by ongoing pain with steady or dysesthetic pain, such as burning or aching, and paroxysmal pain such as shooting or stabbing. In conditions such as diabetic neuropathy, changes in the membrane-bound proteins that form ion channels may alter the electrical properties of the injured neuron, called remodeling. The net effect of membrane remodeling is greater excitability of neurons, leading to a tendency towards action potential generation and propagation in injured primary sensory neurons which occurs in the context of nerve injury and disease. Over the past decade, a new endogenous cannabinoid receptor-mediated system within the nervous system and upon immune-mediated cells has been described. The cannabinoid receptor system consists of two receptors, CB1 and CB2 receptors, as well as endogenously produced endocannabinoids which agonize these receptors.

This is a multicenter trial amongst Western Canadian sites to compare the efficacy of nabilone versus placebo in treating patients with chronic neuropathic pain (NeP) due to diabetic peripheral neuropathy (DPN).

A one-week screening period will occur, during which pain scores and sleep scores will be tabulated. Following screening, a 4-week period of single blind treatment with flexible dosing of nabilone at 0.5 - 4 mg/day will initiate. All subjects will begin with nabilone therapy of 1 mg daily for a minimum of 4 days, with the dose of the study medication assessed and adjusted either upwards or downwards as needed to balance efficacy for pain control with tolerability of possible side effects. All subjects who experience at least a 30% reduction in their weekly mean pain score during the single blind flexible dosing phase will be considered a responder, and will be further continued in the study. During the double-blind portion of the study, subjects randomized to nabilone will continue on the dose of nabilone achieved at the completion of the single-blind phase, and this dose will be maintained throughout the double-blind phase. Subjects randomized to placebo will receive 1 mg of nabilone daily for one week, followed by 4 consecutive weeks of placebo. This dose of nabilone will permit a tapering for those subjects achieving a higher daily dose of nabilone during the single-blind phase, or will maintain those who were taking only 1 mg per day in the single-blind phase, preventing an abrupt termination of treatment in subjects who are randomized into the placebo portion of the study.

DETAILED DESCRIPTION:
This is a multicenter trial amongst 3 Western Canadian sites to compare the efficacy of nabilone versus placebo in treating patients with chronic neuropathic pain (NeP) due to diabetic peripheral neuropathy (DPN).

A one-week screening period will occur, during which pain scores and sleep scores will be tabulated.

Following screening, a 4-week period of single blind treatment with nabilone 0.5 - 4 mg/day flexible dosing will take place. All subjects will begin with nabilone therapy of 1 mg daily for a minimum of 4 days, with the dose of the study medication assessed and adjusted either upwards or downwards as needed to balance efficacy for pain control with tolerability for possible side effects.

All subjects who experience at least a 30% reduction in their weekly mean pain score during the single blind flexible dosing phase will be considered a responder, and will be further continued in the study. Those failing to achieve this level of pain relief will be discontinued from further study. Responders will be randomized to 5 weeks of double-blind treatment with nabilone or placebo. The double-blind phase of this study will permit confirmation of efficacy observed during the single-blind phase of the study. During the double-blind portion of the study, subjects randomized to nabilone will continue on the dose of nabilone achieved at the completion of the single-blind phase, and this dose will be maintained throughout the double-blind phase. Subjects randomized to placebo will receive a direct switch to placebo. All subjects will maintain their pre-study doses of analgesic medication for pain control throughout the study.

There will be four total trial phases:

1. Screening Phase This will consist of a 7-day period of time following Visit 1 in which subjects will be monitored for satisfaction of inclusion/exclusion criteria. If other medications are being used for treatment of peripheral neuropathic pain, then these subjects must be on a stable dose for ≥ 30 days prior to entering the single-blind phase (Visit 2). At the end of this screening phase, subjects who meet all inclusion and exclusion criteria will next enter the single-blind phase.
2. Single Blind Flexible Dose Nabilone Treatment Phase This is a 4 week (28 day) treatment period when subjects will take nabilone in a single-blind fashion, at a dose of 1-4 mg per day. All subjects will start with nabilone 0.5 mg po bid (1 mg daily) for at least 4 days, and then their study medication will be assessed and adjusted upwards, or downwards, as needed to achieve optimal NeP relief as well as side effect tolerability. Dosing adjustments will occur at a maximum of once weekly, with the maximum dose of 4 mg per day preventing any further increase in dose, and a minimum dose of 0.5 mg per day preventing any further decrease in dose. At the end of this single-blind phase, all subjects who are deemed a responder (those who experience a ≥ 30% reduction in weekly mean pain score) will be randomized to the double-blind phase. Those subjects who are not a responder will enter the taper phase of the study, with end of treatment assessments performed. Those patients receiving a dose of 0.5 mg daily will receive a single capsule of 0.5 mg at qhs only. In order to prevent potential unmasking, those patients who are intolerant of placebo will also have their placebo dose reduced from 2 capsules daily to one capsule daily.
3. Double Blind Treatment Phase This is a 5 week (35 day) treatment period where subjects deemed to be a responder during the single blind phase will be randomized to double blind treatment with the dose of nabilone achieved at the last week (Visit 5) of the single-blind phase (the dose which optimized NeP relief with side effect tolerability) or placebo. Subjects will be randomized to 1 of 2 treatment groups in a 1:1 ratio, nabilone or placebo respectively. Those subjects randomized to placebo will be directly switched from active drug to placebo for the duration of the study. All subjects will maintain their pre-study doses of analgesic medication for pain control throughout the study. No further dose adjustments will be allowed during Week 4 onward.
4. Taper Phase This is a one week (7 day) period during which patients will taper off of nabilone. All subjects using nabilone will have their dose adjusted (or continued) as 0.5-1 mg nabilone daily. Any subjects using placebo prior to the taper phase will be continued on placebo during the taper phase.

During the single blind phase, the dose of nabilone may be adjusted upward from 1 to 4 mg/day based on tolerability at weekly visits.. Any upward dose adjustments will occur in increments of either 1 or 2 mg/day (if the initial dose is 1 mg or 2 mg per day respectively). If intolerable adverse events occur during any time of the single blind dose adjustment phase, the dose of nabilone may be decreased by 0.5, 1 or 2 mg/day (if the initial dose is 1 mg, 2 mg or 4 mg per day respectively). A dose of 0.5 mg per day which is not tolerated will lead to study termination. Once a dose reduction has taken place, no further dose adjustments will be permitted. An unscheduled visit between study week 3 and study week 4 will be the last opportunity for dose adjustment.

During the double blind phase, subjects must maintain the same dosing regimen achieved at the end of the single blind dose adjustment phase until the end of Week 8 (Visit 7).

At time of completion of the double blind phase, all subjects taking nabilone will taper off of study medication.

All subjects will be required to attend a minimum of 8 visits in person, with one optional additional visit for dose adjustment permitted during the single blind phase.

There will be a total of 9 clinic visits and 3 telephone interviews. Telephone interviews will occur during weeks in which the subject will not be required to attend clinic. The schedule of visits and telephone interviews is as follows:

* Screening (beginning of Week [-1]) (Visit 1)
* Single Blind Dose Treatment - Day 0 (Visit 2)
* Single Blind Flexible Dose Treatment - Day 7 (Visit 3)
* Single Blind Flexible Dose Treatment - Day 14 (Visit 4)
* Telephone Interview - Day 21
* End of Single Blind Flexible Dose Treatment with Determination of Responders, and possible randomization to Double Blind Phase - Day 28 (Visit 5)
* Double Blind Fixed Dose Treatment - Day 35 (Visit 6)
* Telephone Interview - Day 42
* Double Blind Fixed Dose Treatment - Day 49 (Visit 7)
* Telephone Interview - Day 56
* End of Double Blind Fixed Dose Treatment - Day 63 (Visit 8)
* Follow-up Visit following tapering - Day 70 (Visit 9)

There is an optional dose adjustment period (at the end of Week 3). The necessity of this unscheduled visit is to be determined at the discretion of the investigator and is to be arranged by a telephone contact between the investigator and subject If there are concerns regarding dosing of nabilone, adjustments will be permitted at this time.

If a subject prematurely discontinues the study and stops study drug, the end of treatment assessments will be completed as soon as possible, given continued subject consent.

All investigators will be aware of study design and subject treatment during the single-blind phase of study. It is important that the subject remain blinded to the nature of treatment during all phases of study. The subjects will be treated at all times, as if they were on active treatment of nabilone. If any subject becomes aware of their treatment type during any phase of the study, their participation must be discontinued.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects, ages between 18-80 years;
* Signed and dated informed consent;
* Females of childbearing potential must have a negative serum β-HCG pregnancy test and be practicing an effective form of contraception (accepted methods are hormonal [oral contraceptive or injectable contraceptive], double barrier with spermicide, or intrauterine device-IUD). Complete abstinence may be considered acceptable, but must be determined on a case-by-case basis with the clinical investigator.
* Diagnosis of DPN-associated NeP syndrome, confirmed by a qualified Neurologist or pain specialist, with persistence for a minimum of 3 months.
* Score of ≥4 on the DN4 questionnaire, a single page survey consisting of historical questions and one examination portion using light touch and pinprick over the region of suspected neuropathic pain. This has high sensitivity and specificity for neuropathic pain.
* Must complete ≥4 daily pain diaries during the week of the screening phase prior to randomization;
* Must have a daily mean pain score of ≥4 over the screening period prior to randomization based on Daily Pain Rating Scale (DPRS);
* Must have a score of >40 mm on the visual analog scale (VAS) of the Short Form McGill Pain Questionnaire (SF-MPQ);
* Screening laboratory values must be within normal limits, or abnormalities must be deemed clinically insignificant in the judgment of the investigator
* Subject must be deemed capable of complying with study schedule, procedures and medications.

Exclusion Criteria

* Pregnant or lactating women or women of childbearing potential not using acceptable method of contraception;
* Subjects with neuropathic pain that is not due to DPN
* Any skin conditions in the affected areas with NeP that (in the judgment of the investigator) could interfere with evaluation of the NeP
* Current or past DSM-IV-TRTM (2000) diagnosis of schizophrenia, psychotic disorder, bipolar affective disorder or obsessive-compulsive disorder and Major Depressive Disorder (MDD);
* Current or past DSM-IV-TRTM (2000) diagnosis of substance abuse or dependence within the last 6 month;
* Use of marijuana or other cannabinoids during the study. Discontinuation of these substances 30 days prior to the screening visit is permitted. The study consent must be signed and dated prior to the discontinuation of these substances;
* Clinically significant or unstable conditions that, in the opinion of the investigator, would compromise participation in the study. This includes, for example, medical conditions such as, but not limited to: hepatic, renal, respiratory, hematological, immunologic, or cardiovascular diseases (eg, myocardial infarction within previous month, ventricular arrhythmia recent severe heart insufficiency), inflammatory or rheumatologic disease, active infections, symptomatic peripheral vascular disease, and untreated endocrine disorders;
* History of seizure disorder, except febrile seizures of childhood;
* A glycated hemoglobin (HbA1C) of more than 11% at screening
* Any other condition, which in the investigator's judgment might increase the risk to the subject or decrease the chance of obtaining satisfactory data to achieve the objectives of the study. This includes any condition precluding nabilone use;
* Malignancy within past 2 years with exception of basal cell carcinoma;
* Urine screen positive for illicit substances, including tetrahydrocannaboids (THC) such as marijuana at screening (Visit 1);
* Liver function tests or liver enzymes >3 times the upper limit of normal (ULN)
* Other blood or urine laboratory results which are sufficiently abnormal in the view of the investigator(s) to raise concern about the enrollment of this subject in this study.
* A previous history of intolerance or hypersensitivity to cannabinoids or other medications or substances with similar chemical structure;
* Anticipated need for surgery during the study or within 4 weeks of completion;
* Anticipated need for general anesthetics during the course of the study;
* Anticipated need for hospitalization for any reason during the course of the study or within 4 weeks of completion;
* Previous prescribed use of nabilone or other cannabinoids, including use of sample medications, within the 30 days prior to screening. Note that prior use of marijuana is not an exclusion criterion.
* Participation in any other studies involving investigational or marketed products, concomitantly or within 30 days prior to entry in the study and/or
* Employees or relatives of employees of the investigational site or Valeant Canada

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of nabilone compared to placebo in the treatment of diabetic neuropathy-associated peripheral neuropathic pain (DPN). | 2008 - 2012

SECONDARY OUTCOMES:
To evaluate safety and tolerability of nabilone for the treatment of neuropathic pain in subjects with diabetic peripheral neuropathy. | 2008 - 2012

CONTACTS AND LOCATIONS:
Overall Officials: Cory Toth, MD, Principal Investigator — U of Calgary
Locations (1):
- Hotchkiss Brain Institute, Calgary, Alberta, Canada